CLINICAL TRIAL: NCT05496894
Title: A Phase Ⅱ Study to Evaluate the Safety and Efficacy of Mitoxantrone Hydrochloride Liposome Injection for Relapsing Multiple Sclerosis
Brief Title: A Study of Mitoxantrone Hydrochloride Liposome Injection for Relapsing Multiple Sclerosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the company's project adjustment, decided to stop this study
Sponsor: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE071-CSP-030
Record Dates: First submitted 2022-07-28; First posted 2022-08-11 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Relapsing Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mitoxantrone Hydrochloride Liposome Injection 4 mg/m^2 group (Experimental): Participants will receive Mitoxantrone Hydrochloride Liposome Injection 4 mg/m^2 every 3 months (Q3M).
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome Injection
- Mitoxantrone Hydrochloride Liposome Injection 8 mg/m^2 group (Experimental): Participants will receive Mitoxantrone Hydrochloride Liposome Injection 8 mg/m^2 every 3 months (Q3M).
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome Injection
- Mitoxantrone Hydrochloride Liposome Injection 12 mg/m^2 group (Experimental): Participants will receive Mitoxantrone Hydrochloride Liposome Injection 12 mg/m^2 every 3 months (Q3M).
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome Injection

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome Injection — IV, once every 3 months (Q3M)

SUMMARY:
This is a multicenter, randomized, single-arm, open-label Phase II study to evaluate the efficacy and safety of Mitoxantrone Hydrochloride Liposome Injection with different doses in participants with Relapsing Multiple Sclerosis. Participants will be randomly enrolled into three treatment groups: Mitoxantrone Hydrochloride Liposome Injection 4 mg/m^2 group, Mitoxantrone Hydrochloride Liposome Injection 8 mg/m^2 group, and Mitoxantrone Hydrochloride Liposome Injection 12 mg/m^2 group. The primary outcome measure is the cumulative number of new Gd-enhancing lesions at the end of 48 weeks of Mitoxantrone Hydrochloride Liposome Injection treatment in brain MRI.

DETAILED DESCRIPTION:
Multiple sclerosis is a chronic, inflammatory, demyelinating disease of the central nervous system (CNS) and is one of the most common causes of neurological disability in young adults. It is characterised by multi-focal recurrent attacks of neurological symptoms and signs with variable recovery.This is a multicenter, randomized, single-arm, open-label Phase II study to evaluate the efficacy and safety of Mitoxantrone Hydrochloride Liposome Injection with different doses in participants with Relapsing Multiple Sclerosis. Participants will be randomly enrolled into three treatment groups: Mitoxantrone Hydrochloride Liposome Injection 4 mg/m^2 group, Mitoxantrone Hydrochloride Liposome Injection 8 mg/m^2 group, and Mitoxantrone Hydrochloride Liposome Injection 12 mg/m^2 group. The primary outcome measure is the cumulative number of new Gd-enhancing lesions at the end of 48 weeks of Mitoxantrone Hydrochloride Liposome Injection treatment in brain MRI.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 55 years of age (inclusive);
* Diagnosis of relapsing multiple sclerosis (RMS);
* Disease duration of secondary progressive multiple sclerosis (SPMS) with superimposed relapses ≤ 5 years;
* Expanded disability status scale (EDSS) score of 3 to 8;
* Participants who have received disease-modifying therapy still relapse or aggravate; or participants who, in the opinion of the investigator, are suitable for treatment with Mitoxantrone Hydrochloride Liposome Injection;
* Participants voluntarily sign informed consent, and complete the study according to the protocol.

Exclusion Criteria:

* Pregnant or lactating female participants or participants planning to have a child during the study;
* History of severe drug allergy, or allergy or intolerance to gadolinium, anthracyclines or liposome drugs;
* History of vitamin B12 deficiency;
* Participants with malignant tumor diagnosed within 5 years before the screening phase, except the skin basal cell carcinoma under effective control, and Stage I Squamous Cell Carcinoma);
* Participants with history of interstitial lung disease or with pneumonia according to chest X-ray in the screening phase;
* Participants with serious or active skin diseases, or clinically significant skin abnormalities in physical examination in the screening phase;
* History of severe immunodeficiency;
* History of drug and/or alcohol abuse, or mental disorder;
* Participants has a progressive neurological disorder or optic neuritis other than MS; or has other disease that should be treated more preferentially than MS, or that could interfere with the study or compromise participants compliance with treatment;
* MRI before randomization shows cervical spinal cord compression or lesions in non-MS characteristic areas of the brain, and the lesions can explain the changes in clinical symptoms and signs;
* MS relapse in the screening phase;
* Participated in other drug clinical studies and received investigational product within 3 months before screening or within 5 half-lives of the investigational product (whichever was longer), or participated in medical device clinical studies which is judged by the investigator to have a possible impact on the results of this study;
* Participants who have received disease-modifying therapy or immunosuppressive agents or systemic corticosteroids within the washout period before the first dose (e.g., 4 weeks for interferon, PEGylated interferon, glatiramer acetate, dimethyl fumarate and 12 weeks for fingolimod, siponimod, intravenous immunoglobulin or plasma exchange, etc.)
* Participants who have received anthracyclines or cardiotoxic drugs before screening;
* Participants who previously received total body irradiation or total lymphatic irradiation, or received stem cell therapy or any type of bone marrow transplantation, or received solid organ transplantation;
* Presence of the following clinically significant diseases: myocardial infarction, acute coronary syndrome, viral myocarditis, pulmonary embolism within 6 months; coronary revascularization within 6 months; arrhythmia requiring Class Ia or Ш antiarrhythmic drugs;
* Laboratory tests in screening phase, such as white blood cell count, neutrophil count, platelet count, hemoglobin, creatinine clearance, etc., are abnormal with clinical significance (according to the judgment of the investigator); positive results for Hepatitis B Surface Antigen (HBsAg), Hepatitis C Antibody (HCVAb), syphilis antibody test; total bilirubin > 1.5x ULN, or alanine aminotransferase or aspartate aminotransferase > 3x ULN;
* Participants could not complete MRI scan before randomization, such as participants with claustrophobia;
* Participants with active or uncontrolled infection (defined as requiring systemic anti-infective therapy and the temperature ≥ 38℃ (axillary temperature) before receiving drugs and unexplainable);
* Investigator believe that participants have other disease that are not suitable for participating in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
The cumulative number of new Gadolinium (Gd)-enhancing lesions at the end of 48 weeks of Mitoxantrone Hydrochloride Liposome Injection treatment in brain MRI. | Week 48

SECONDARY OUTCOMES:
Annualized Relapse Rate (ARR) | Week 48
  ARR at Week 48 is calculated as the ratio of the sum of all participants confirmed relapse counts divided by the sum of all participants treatment duration (in years).
Number of Relapses | Week 48
Time to Onset of Confirmed Disability Progression for at least 6 Months | Week 48
Time to Onset of Confirmed Disability Progression for at least 3 Months | Week 48
Proportion of participants with ≥ 20% improvement from baseline in T25FW walking speed. | Week 48
Change from baseline to Week 48 in T25FW walking speed. | Week 48
Number of new or enlarged T2 lesions. | Week 48
Change from baseline in brain MRI Gd-enhancing T1 lesion volume at Weeks 12、24、36、48. | Week 12、24、36、48
Change from baseline in brain MRI T2 lesion volume at Weeks 12、24、36、48. | Week 12、24、36、48
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Week 56
Plasma concentration of Mitoxantrone Hydrochloride Liposome Injection. | Week 12
Descriptive analysis of the rate of change in the number or proportion of B cells from baseline to different time points in different dose groups. | Week 36
Descriptive analysis of the rate of change in the number or proportion of T cells from baseline to different time points in different dose groups. | Week 36
Descriptive analysis of the rate of change in the number or proportion of NK cells from baseline to different time points in different dose groups. | Week 36

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No